CLINICAL TRIAL: NCT03858452
Title: Evaluation of Functional Relations and Their Changes Between Pelvic Floor, Diaphragm and Trunk Muscles in Men After Radical Prostatectomy
Brief Title: Relations Between Pelvic Floor, Diaphragm and Trunk Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Zemyna Milasauskiene, Head of Research and Studies Coordination Centre, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BE-2-61
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer; Urinary Incontinence
Keywords: Prostatectomy; Rehabilitation; Incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pelvic floor muscles training group (Active Comparator): Pelvic floor muscles exercises twice a day for 30 min
  Interventions: Procedure: Muscles exercises program
- Diaphragm muscles training group (Active Comparator): Breathing exercises twice a day for 30 min
  Interventions: Procedure: Muscles exercises program
- Abdominal muscles training group (Active Comparator): Abdominal muscles exercises twice a day for 30 min
  Interventions: Procedure: Muscles exercises program

INTERVENTIONS:
Procedure: Muscles exercises program

SUMMARY:
The present study evaluates the functional relations of pelvic floor, diaphragm, and torso muscles, their variation and correlations with urinary incontinence while separately training physical characteristics of the mentioned muscles in men after radical prostatectomy.

DETAILED DESCRIPTION:
During the last two decades, the connection between pelvic floor muscles (PFM) and abdominal muscles or diaphragm has been detected: PFM contract and relax during the inhalation and exhalation in pace with the diaphragm; the activity of the PFM increases with the increase of intra-abdominal pressure during forced exhalations or cough. The role of pelvic floor is essential for the synergy of diaphragm and abdominal muscles in maintenance of intra-abdominal pressure. According to the aforementioned physiological functional relationships, the investigators have postulated a hypothesis that diaphragm muscles training and abdominal muscles training could have similar effect as direct PFM training on pelvic floor muscles strength and pelvic floor muscles endurance measured using perineometer in men after radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* stable somatic state
* written informed consent.

Exclusion Criteria:

* chronic obstructive pulmonary disease,
* surgical interventions in abdominal area,
* complains in lower back,
* acute musculoskeletal injuries in last 6 months
* cognitive dysfunction

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2012-05-30 (Actual); Study Completion 2012-12-30 (Actual)

PRIMARY OUTCOMES:
Effect of activation of different muscles groups on pelvic floor muscles strength | 6 months after radical prostatectomy.
  Pelvic floor muscles strength was measured in cmH2O
Effect of activation of different muscles groups on pelvic floor muscles endurance. | 6 months after radical prostatectomy.
  Pelvic floor muscles endurance was measured in seconds.

SECONDARY OUTCOMES:
Urinary loss dynamics | 6 month after radical prostatectomy
  Pad weight by grams during 8 hours pad test
correlation between urinary incontinence and pelvic floor muscles strength and endurance dynamics | 6 months after radical prostatectomy
  correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Daimantas Milonas, MD, PhD, Principal Investigator — LUHS

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Data access request will be reviewed by investigators. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Result] Zachovajeviene B, Siupsinskas L, Zachovajevas P, Milonas D. Dynamics of pelvic floor muscle functional parameters and their correlations with urinary incontinence in men after radical prostatectomy. Neurourol Urodyn. 2017 Jan;36(1):126-131. doi: 10.1002/nau.22887. Epub 2015 Sep 30. PMID 26421383